CLINICAL TRIAL: NCT06650930
Title: Pharmacokinetics of Oral Calcium Carbonate in Parturients
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jessica Ansari, MD, MS, Principal Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 77182
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Pregnancy; Pharmacokinetics; Postpartum Hemorrhage
Keywords: calcium; oral calcium; calcium carbonate; calcium pharmacokinetics; pharmacokinetics in pregnancy; postpartum hemorrhage; ionized calcium; pharmacokinetics
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Calcium Carbonate

STUDY DESIGN:
Intervention Model Description: This is a single arm pharmacokinetic trial. No efficacy outcomes are analyzed. The aim of the study is to determine the pharmacokinetics of a single dose of oral calcium carbonate in parturients. The outcome of interest is serial measurement of the ionized calcium in the blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oral calcium carbonate (Experimental): Patients take a single dose of oral calcium carbonate 3000mg
  Interventions: Drug: Oral calcium carbonate

INTERVENTIONS:
Drug: Oral calcium carbonate — All participants receive a single, open-label dose of oral calcium carbonate 3000mg

SUMMARY:
This study investigates the time course of change in calcium in the blood after a pregnant subject takes an oral dose of calcium carbonate (commonly marketed as "Tums"). This information is important for trials investigating whether calcium can reduce postpartum hemorrhage, bleeding after delivery.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant female subjects at the study institution, admitted for labor (spontaneous, augmented, or induced)

Exclusion Criteria:

1. severe range blood pressure (BP >160/>110) within the 48 hours prior to delivery
2. patient age <18 years or >45 years
3. renal dysfunction with a documented serum Cr > 1.0 mg/dL
4. known history of congenital or acquired cardiac disease or history of arrhythmia
5. patient taking digoxin
6. patient currently taking a calcium channel blocker
7. Weight <55kg or >100kg, or
8. receiving magnesium infusion within 24 hours prior to or during cesarean delivery
9. Prior or planned administration of calcium by the obstetric or anesthesiology teams for clinical indications within 24 hours of study enrollment
10. Patient took a calcium supplement in the past 48 hours
11. Patient status is NPO (nothing by mouth) as ordered by the clinical team

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Ionized calcium concentration | 4 hours
  Ionized calcium (mmol/L) is measured at baseline and over 5 additional convenience timepoints over the 4 hours after ingestion of calcium carbonate 3000mg.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Ansari, MD, MS, Principal Investigator — Stanford University
Locations (1):
- Stanford Children's Health, Lucile Packard Children's Hospital, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
Patient privacy

REFERENCES:
- [Background] Ansari JR, Yarmosh A, Michel G, Lyell D, Hedlin H, Cornfield DN, Carvalho B, Bateman BT. Intravenous Calcium to Decrease Blood Loss During Intrapartum Cesarean Delivery: A Randomized Controlled Trial. Obstet Gynecol. 2024 Jan 1;143(1):104-112. doi: 10.1097/AOG.0000000000005441. Epub 2023 Nov 3. PMID 37917943
- [Background] Ansari JR, Kalariya N, Carvalho B, Flood P, Guo N, Riley E. Calcium chloride for the prevention of uterine atony during cesarean delivery: A pilot randomized controlled trial and pharmacokinetic study. J Clin Anesth. 2022 Sep;80:110796. doi: 10.1016/j.jclinane.2022.110796. Epub 2022 Apr 18. PMID 35447502
- [Background] Ansari JR, Conti DJ, Michel G, Yarmosh A, Cole NM, Shafer SL. Bioequivalence and Pharmacokinetics of Intravenous Calcium during Cesarean Delivery. Anesthesiology. 2025 Jan 1;142(1):121-131. doi: 10.1097/ALN.0000000000005248. PMID 39361822
- [Background] Ansari J, Carvalho B, Shafer SL, Flood P. Pharmacokinetics and Pharmacodynamics of Drugs Commonly Used in Pregnancy and Parturition. Anesth Analg. 2016 Mar;122(3):786-804. doi: 10.1213/ANE.0000000000001143. PMID 26891392